CLINICAL TRIAL: NCT05863949
Title: STOP Vertigo: Supplementation of Vitamin D for Termination of Recurrences From Benign Paroxysmal Positional Vertigo
Brief Title: Clinical Trial of Vit D and Calcium for Recurrent BPPV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Darren Tse, Physician, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20220451-01T
Record Dates: First submitted 2023-04-28; First posted 2023-05-18 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: BPPV; Benign Paroxysmal Positional Vertigo; Vertigo; Vertigo, Peripheral; Dizziness; Dizziness; Epidemic; Vitamin D Deficiency; Calcium Deficiency
Keywords: bppv; benign paroxysmal positional vertigo; vertigo; dizziness; vitamin D
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo; Dizziness; Vitamin D Deficiency | interventions — S100 Calcium Binding Protein G

STUDY DESIGN:
Intervention Model Description: This is an off-label, multicenter, randomized, clinical trial in vitamin D deficient adults aged 18 and above with recurrent BPPV. Its goal is to determine whether vitamin D supplementation, with or without calcium supplementation, compared with placebo will decrease the frequency of recurrent episodes of BPPV. A total of 860 vitamin D deficient adults diagnosed with recurrent BPPV will be enrolled at participating clinical study sites.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Enrolled subjects will be blinded to their treatment assignment. Both study staff and trial investigators will be blinded to treatment assignments and will remain blinded throughout the course of the trial. Randomization (treatment assignment) will be performed via computer algorithm based on subject ID. Randomization codes will be maintained in a password protected, encrypted file available only to the single unmasked investigator at each site, in order to prevent accidental unmasking of other trial personnel. All care will be taken to ensure that the study team are kept blinded.
  Pills, which will be dispensed at 3-month intervals, will be indistinguishable between groups. They will be dispensed in kits that are labeled as outlined in section 6.2 Study Drug Packaging and Labeling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vitamin D +/- calcium supplementation (Experimental): patients given Vitamin D 1000iu daily. Also given calcium 500mg BID daily if calcium deficient.
  Interventions: Dietary Supplement: vitamin D +/- calcium
- Placebo arm (Placebo Comparator): patients given 3 pills of placebo daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: vitamin D +/- calcium — vitamin D 1000iU daily +/- calcium 500mg BID daily
  Arms: vitamin D +/- calcium supplementation
Other: Placebo — placebo pill x3 daily
  Arms: Placebo arm

SUMMARY:
Randomized double blind placebo controlled trial of vitamin D supplements, with or without calcium supplementation, versus placebo in reduction of recurrences in BPPV.

DETAILED DESCRIPTION:
Benign paroxysmal positional vertigo (BPPV) is the most common neuro-otological disorder, with a lifetime prevalence of 2.4 percent.1 BPPV is responsible for nearly one-half of cases of peripheral vestibular dysfunction. It is a highly recurrent disorder, with more than 1 in 4 patients experiencing a second attack, often within 6 months of the first.2-4 According to the Clinical Practice Guidelines for BPPV from the American Academy of Otolaryngology-Head and Neck Surgery Foundation, particle repositioning maneuvers (PRMs) are the only recommended treatment to resolve symptoms for both initial BPPV episodes as well as persistent episodes.5 While attacks can be effectively treated by PRMs, these often must be performed by a physician or other trained healthcare professional, and sometimes multiple attempts are required in order to successfully resolve a patient's symptoms. Furthermore, even with effective particle repositioning, a subset of patients may continue to experience bouts of recurrent attacks, up to several times yearly. The attacks themselves, as well as the nature of their treatment, - especially in patients with recurrent episodes - are prone to lead to interruptions in patients' daily activities, cause sick leaves, and result in significant direct and indirect costs to both the patient and the healthcare system.6 The prevalence of BPPV increases with age and elderly patients with BPPV are more likely to have reduced activities of daily living (ADL) scores, sustain falls, and suffer from depression.4,7 In the United States (US), more than sixty-five percent of patients with BPPV experience potentially avoidable diagnostic testing or therapeutic interventions during the time leading up to a proper diagnosis, costing the US health care system nearly $2 billion per year.5

BPPV is widely accepted to be caused by otoconia that are dislodged from the utricular macula into the semicircular canals - most commonly the posterior canal.8 Otoconia are made of a largely organic core of glycoproteins, with a predominantly inorganic periphery of calcium carbonate.9 Otoconia form within the otherwise low-calcium endolymph via an active, tightly controlled and ordered process.10 Recent studies have shown that the biomineralization of otoconia has similarities to that of bone and teeth, and that bone metabolism has a connection to BPPV. 11-13 Furthermore, an association has been demonstrated between BPPV and osteoporosis, and otoconia formation has been shown to be dysfunctional in animal models of osteoporosis.14,15

The impact of recurrent BPPV on both patients and the healthcare system is multiplicative. With each episode of recurrence, patients become symptomatic - potentially severely so - and must seek treatment again in the form of particle repositioning maneuvers. These patients therefore suffer further functional impairment, potentially missed school and work, and require healthcare interventions which are not without cost to the system. No preventative treatment option for recurrent BPPV exists. Establishing such a preventative treatment would have significant implications in reducing both direct and indirect costs of this highly prevalent and recurrent disorder.

Vitamin D is involved in bodily calcium regulation, and thus poses an attractive potential treatment for BPPV. Vitamin D deficiency is common in many regions worldwide, and supplementation carries little risk. A body of literature has emerged to date investigating potential links between vitamin D deficiency and BPPV - especially recurrent - and whether vitamin D supplementation could in turn serve some role in treatment or prevention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* 2 or more distinct episodes of benign paroxysmal positional vertigo within a 12-month period on history
* At least 1 episode diagnosed based on physical examination by trained study personnel, meeting the diagnostic criteria of the Bárány Society
* Episodes separated in time, with a minimum of 1 week symptom-free between episodes
* Serum evidence of Vitamin D deficiency, as evidenced by 25-hydroxy vitamin D level of <75 nmol/L (<30 ng/mL)48
* Subject able to provide informed consent to participate in the study

Exclusion Criteria:

Potential subjects will be excluded if they

* have another identifiable cause of vertigo identified on history or physical examination
* have a history of allergy or medically significant adverse reaction to vitamin D or calcium carbonate
* have a chronic medical disorder which is a contraindication to vitamin D or calcium carbonate supplementation, including uncontrolled hyperparathyroidism, nephrolithiasis, or GI malabsorption disorders
* are on loop diuretic agents or thiazides
* have a contraindication to routine bloodwork for study purposes, including being hospitalized with a critical illness, cellulitis at blood draw sites, or presence of vascular grafts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of BPPV | 1 year
  how many recurrences of BPPV

SECONDARY OUTCOMES:
serum vitamin D levels (25(OH)D3) | 1 year
  serum vitamin D levels
proportion of serum vitamin D normalization | 1 year
  do patients normalize
time to serum vitamin D normalization | 1 year
  how long does it take patients to normalize
proportion of recurrences | 1 year
  what proportion of total patients have recurrences
duration of recurrences | 1 year
  how long do recurrences of BPPV last
EQ-5D | 1 year
  quality of life measurement
days per year of missed school/work | 1 year
  days per year of missed school/work

CONTACTS AND LOCATIONS:
Overall Officials: Darren Tse, MD, Principal Investigator — Ottawa Hospita Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] von Brevern M, Bertholon P, Brandt T, Fife T, Imai T, Nuti D, Newman-Toker D. Benign paroxysmal positional vertigo: Diagnostic criteria. J Vestib Res. 2015;25(3-4):105-17. doi: 10.3233/VES-150553. PMID 26756126
- [Background] Luryi AL, Lawrence J, Bojrab DI, LaRouere M, Babu S, Zappia J, Sargent EW, Chan E, Naumann I, Hong RS, Schutt CA. Recurrence in Benign Paroxysmal Positional Vertigo: A Large, Single-Institution Study. Otol Neurotol. 2018 Jun;39(5):622-627. doi: 10.1097/MAO.0000000000001800. PMID 29649052
- [Background] Perez P, Franco V, Cuesta P, Aldama P, Alvarez MJ, Mendez JC. Recurrence of benign paroxysmal positional vertigo. Otol Neurotol. 2012 Apr;33(3):437-43. doi: 10.1097/MAO.0b013e3182487f78. PMID 22388730
- [Background] Zhu CT, Zhao XQ, Ju Y, Wang Y, Chen MM, Cui Y. Clinical Characteristics and Risk Factors for the Recurrence of Benign Paroxysmal Positional Vertigo. Front Neurol. 2019 Nov 13;10:1190. doi: 10.3389/fneur.2019.01190. eCollection 2019. PMID 31798518
- [Background] Bhattacharyya N, Gubbels SP, Schwartz SR, Edlow JA, El-Kashlan H, Fife T, Holmberg JM, Mahoney K, Hollingsworth DB, Roberts R, Seidman MD, Steiner RW, Do BT, Voelker CC, Waguespack RW, Corrigan MD. Clinical Practice Guideline: Benign Paroxysmal Positional Vertigo (Update). Otolaryngol Head Neck Surg. 2017 Mar;156(3_suppl):S1-S47. doi: 10.1177/0194599816689667. PMID 28248609
- [Background] von Brevern M, Radtke A, Lezius F, Feldmann M, Ziese T, Lempert T, Neuhauser H. Epidemiology of benign paroxysmal positional vertigo: a population based study. J Neurol Neurosurg Psychiatry. 2007 Jul;78(7):710-5. doi: 10.1136/jnnp.2006.100420. Epub 2006 Nov 29. PMID 17135456
- [Background] Oghalai JS, Manolidis S, Barth JL, Stewart MG, Jenkins HA. Unrecognized benign paroxysmal positional vertigo in elderly patients. Otolaryngol Head Neck Surg. 2000 May;122(5):630-4. doi: 10.1016/S0194-5998(00)70187-2. PMID 10793337
- [Background] Parnes LS, Agrawal SK, Atlas J. Diagnosis and management of benign paroxysmal positional vertigo (BPPV). CMAJ. 2003 Sep 30;169(7):681-93. PMID 14517129
- [Background] Lins U, Farina M, Kurc M, Riordan G, Thalmann R, Thalmann I, Kachar B. The otoconia of the guinea pig utricle: internal structure, surface exposure, and interactions with the filament matrix. J Struct Biol. 2000 Jul;131(1):67-78. doi: 10.1006/jsbi.2000.4260. PMID 10945971
- [Background] Lundberg YW, Zhao X, Yamoah EN. Assembly of the otoconia complex to the macular sensory epithelium of the vestibule. Brain Res. 2006 May 26;1091(1):47-57. doi: 10.1016/j.brainres.2006.02.083. Epub 2006 Apr 4. PMID 16600187
- [Background] Zhao X, Yang H, Yamoah EN, Lundberg YW. Gene targeting reveals the role of Oc90 as the essential organizer of the otoconial organic matrix. Dev Biol. 2007 Apr 15;304(2):508-24. doi: 10.1016/j.ydbio.2007.01.013. Epub 2007 Jan 12. PMID 17300776
- [Background] Xu Y, Zhang H, Yang H, Zhao X, Lovas S, Lundberg YW. Expression, functional, and structural analysis of proteins critical for otoconia development. Dev Dyn. 2010 Oct;239(10):2659-73. doi: 10.1002/dvdy.22405. PMID 20803598
- [Background] Jeong SH, Choi SH, Kim JY, Koo JW, Kim HJ, Kim JS. Osteopenia and osteoporosis in idiopathic benign positional vertigo. Neurology. 2009 Mar 24;72(12):1069-76. doi: 10.1212/01.wnl.0000345016.33983.e0. PMID 19307540
- [Background] Vibert D, Kompis M, Hausler R. Benign paroxysmal positional vertigo in older women may be related to osteoporosis and osteopenia. Ann Otol Rhinol Laryngol. 2003 Oct;112(10):885-9. doi: 10.1177/000348940311201010. PMID 14587980
- [Background] Vibert D, Sans A, Kompis M, Travo C, Muhlbauer RC, Tschudi I, Boukhaddaoui H, Hausler R. Ultrastructural changes in otoconia of osteoporotic rats. Audiol Neurootol. 2008;13(5):293-301. doi: 10.1159/000124277. Epub 2008 Apr 7. PMID 18391565
- [Background] Yang B, Lu Y, Xing D, Zhong W, Tang Q, Liu J, Yang X. Association between serum vitamin D levels and benign paroxysmal positional vertigo: a systematic review and meta-analysis of observational studies. Eur Arch Otorhinolaryngol. 2020 Jan;277(1):169-177. doi: 10.1007/s00405-019-05694-0. Epub 2019 Oct 19. PMID 31630244
- [Background] Jeong SH, Lee SU, Kim JS. Prevention of recurrent benign paroxysmal positional vertigo with vitamin D supplementation: a meta-analysis. J Neurol. 2022 Feb;269(2):619-626. doi: 10.1007/s00415-020-09952-8. Epub 2020 Aug 7. PMID 32767116
- [Background] Buki B, Ecker M, Junger H, Lundberg YW. Vitamin D deficiency and benign paroxysmal positioning vertigo. Med Hypotheses. 2013 Feb;80(2):201-4. doi: 10.1016/j.mehy.2012.11.029. Epub 2012 Dec 14. PMID 23245911
- [Background] Sheikhzadeh M, Lotfi Y, Mousavi A, Heidari B, Monadi M, Bakhshi E. Influence of supplemental vitamin D on intensity of benign paroxysmal positional vertigo: A longitudinal clinical study. Caspian J Intern Med. 2016 Spring;7(2):93-8. PMID 27386060
- [Background] Talaat HS, Kabel AM, Khaliel LH, Abuhadied G, El-Naga HA, Talaat AS. Reduction of recurrence rate of benign paroxysmal positional vertigo by treatment of severe vitamin D deficiency. Auris Nasus Larynx. 2016 Jun;43(3):237-41. doi: 10.1016/j.anl.2015.08.009. Epub 2015 Sep 16. PMID 26386496
- [Background] Jeong SH, Kim JS, Kim HJ, Choi JY, Koo JW, Choi KD, Park JY, Lee SH, Choi SY, Oh SY, Yang TH, Park JH, Jung I, Ahn S, Kim S. Prevention of benign paroxysmal positional vertigo with vitamin D supplementation: A randomized trial. Neurology. 2020 Sep 1;95(9):e1117-e1125. doi: 10.1212/WNL.0000000000010343. Epub 2020 Aug 5. PMID 32759193
- [Background] Sterne JA, Hernan MA, Reeves BC, Savovic J, Berkman ND, Viswanathan M, Henry D, Altman DG, Ansari MT, Boutron I, Carpenter JR, Chan AW, Churchill R, Deeks JJ, Hrobjartsson A, Kirkham J, Juni P, Loke YK, Pigott TD, Ramsay CR, Regidor D, Rothstein HR, Sandhu L, Santaguida PL, Schunemann HJ, Shea B, Shrier I, Tugwell P, Turner L, Valentine JC, Waddington H, Waters E, Wells GA, Whiting PF, Higgins JP. ROBINS-I: a tool for assessing risk of bias in non-randomised studies of interventions. BMJ. 2016 Oct 12;355:i4919. doi: 10.1136/bmj.i4919. PMID 27733354
- [Background] Mithal A, Wahl DA, Bonjour JP, Burckhardt P, Dawson-Hughes B, Eisman JA, El-Hajj Fuleihan G, Josse RG, Lips P, Morales-Torres J; IOF Committee of Scientific Advisors (CSA) Nutrition Working Group. Global vitamin D status and determinants of hypovitaminosis D. Osteoporos Int. 2009 Nov;20(11):1807-20. doi: 10.1007/s00198-009-0954-6. Epub 2009 Jun 19. PMID 19543765
- [Background] Hagenau T, Vest R, Gissel TN, Poulsen CS, Erlandsen M, Mosekilde L, Vestergaard P. Global vitamin D levels in relation to age, gender, skin pigmentation and latitude: an ecologic meta-regression analysis. Osteoporos Int. 2009 Jan;20(1):133-40. doi: 10.1007/s00198-008-0626-y. Epub 2008 May 6. PMID 18458986
- [Background] Parva NR, Tadepalli S, Singh P, Qian A, Joshi R, Kandala H, Nookala VK, Cheriyath P. Prevalence of Vitamin D Deficiency and Associated Risk Factors in the US Population (2011-2012). Cureus. 2018 Jun 5;10(6):e2741. doi: 10.7759/cureus.2741. PMID 30087817
- [Background] Hanley DA, Davison KS. Vitamin D insufficiency in North America. J Nutr. 2005 Feb;135(2):332-7. doi: 10.1093/jn/135.2.332. PMID 15671237
- [Background] Bischoff-Ferrari HA, Shao A, Dawson-Hughes B, Hathcock J, Giovannucci E, Willett WC. Benefit-risk assessment of vitamin D supplementation. Osteoporos Int. 2010 Jul;21(7):1121-32. doi: 10.1007/s00198-009-1119-3. Epub 2009 Dec 3. PMID 19957164
- [Background] Bjelakovic G, Gluud LL, Nikolova D, Whitfield K, Krstic G, Wetterslev J, Gluud C. Vitamin D supplementation for prevention of cancer in adults. Cochrane Database Syst Rev. 2014 Jun 23;2014(6):CD007469. doi: 10.1002/14651858.CD007469.pub2. PMID 24953955
- [Background] Avenell A, Mak JC, O'Connell D. Vitamin D and vitamin D analogues for preventing fractures in post-menopausal women and older men. Cochrane Database Syst Rev. 2014 Apr 14;2014(4):CD000227. doi: 10.1002/14651858.CD000227.pub4. PMID 24729336
- [Background] Malihi Z, Wu Z, Stewart AW, Lawes CM, Scragg R. Hypercalcemia, hypercalciuria, and kidney stones in long-term studies of vitamin D supplementation: a systematic review and meta-analysis. Am J Clin Nutr. 2016 Oct;104(4):1039-1051. doi: 10.3945/ajcn.116.134981. Epub 2016 Sep 7. PMID 27604776
- [Background] Reid IR. Efficacy, effectiveness and side effects of medications used to prevent fractures. J Intern Med. 2015 Jun;277(6):690-706. doi: 10.1111/joim.12339. PMID 25495429
- [Background] Brazier M, Grados F, Kamel S, Mathieu M, Morel A, Maamer M, Sebert JL, Fardellone P. Clinical and laboratory safety of one year's use of a combination calcium + vitamin D tablet in ambulatory elderly women with vitamin D insufficiency: results of a multicenter, randomized, double-blind, placebo-controlled study. Clin Ther. 2005 Dec;27(12):1885-93. doi: 10.1016/j.clinthera.2005.12.010. PMID 16507374
- [Background] Lewis JR, Zhu K, Prince RL. Adverse events from calcium supplementation: relationship to errors in myocardial infarction self-reporting in randomized controlled trials of calcium supplementation. J Bone Miner Res. 2012 Mar;27(3):719-22. doi: 10.1002/jbmr.1484. PMID 22139587
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Jones G. Pharmacokinetics of vitamin D toxicity. Am J Clin Nutr. 2008 Aug;88(2):582S-586S. doi: 10.1093/ajcn/88.2.582S. PMID 18689406
- [Background] Gallagher JC, Smith LM, Yalamanchili V. Incidence of hypercalciuria and hypercalcemia during vitamin D and calcium supplementation in older women. Menopause. 2014 Nov;21(11):1173-80. doi: 10.1097/GME.0000000000000270. PMID 24937025
- [Background] Kaptchuk TJ, Kelley JM, Conboy LA, Davis RB, Kerr CE, Jacobson EE, Kirsch I, Schyner RN, Nam BH, Nguyen LT, Park M, Rivers AL, McManus C, Kokkotou E, Drossman DA, Goldman P, Lembo AJ. Components of placebo effect: randomised controlled trial in patients with irritable bowel syndrome. BMJ. 2008 May 3;336(7651):999-1003. doi: 10.1136/bmj.39524.439618.25. Epub 2008 Apr 3. PMID 18390493
- [Background] Hrobjartsson A, Gotzsche PC. Placebo interventions for all clinical conditions. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD003974. doi: 10.1002/14651858.CD003974.pub3. PMID 20091554
- [Background] Kaptchuk TJ. Powerful placebo: the dark side of the randomised controlled trial. Lancet. 1998 Jun 6;351(9117):1722-5. doi: 10.1016/S0140-6736(97)10111-8. No abstract available. PMID 9734904
- [Background] Miller FG, Kaptchuk TJ. The power of context: reconceptualizing the placebo effect. J R Soc Med. 2008 May;101(5):222-5. doi: 10.1258/jrsm.2008.070466. No abstract available. PMID 18463276
- [Background] Hrobjartsson A. What are the main methodological problems in the estimation of placebo effects? J Clin Epidemiol. 2002 May;55(5):430-5. doi: 10.1016/s0895-4356(01)00496-6. PMID 12007544
- [Background] Amrein K, Scherkl M, Hoffmann M, Neuwersch-Sommeregger S, Kostenberger M, Tmava Berisha A, Martucci G, Pilz S, Malle O. Vitamin D deficiency 2.0: an update on the current status worldwide. Eur J Clin Nutr. 2020 Nov;74(11):1498-1513. doi: 10.1038/s41430-020-0558-y. Epub 2020 Jan 20. PMID 31959942
- [Background] Pietras SM, Obayan BK, Cai MH, Holick MF. Vitamin D2 treatment for vitamin D deficiency and insufficiency for up to 6 years. Arch Intern Med. 2009 Oct 26;169(19):1806-8. doi: 10.1001/archinternmed.2009.361. No abstract available. PMID 19858440